CLINICAL TRIAL: NCT05337696
Title: Circumferential Vertebral Reconstruction of Osteoporotic Compression Fractures Using a Novel Bipedicular Peek Implant
Acronym: RECONSTRUCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: financial constraints
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Tomoyoshi Shigematsu, Assistant Professor, Neurosurgery, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01269
Record Dates: First submitted 2022-03-26; First posted 2022-04-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Vertebral Compression Fractures; Osteoporotic Vertebral Compression Fractures
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participants with vertebral compression fractures (Experimental): Participants with vertebral compression fractures who have failed conservative care strategies.
  Interventions: Procedure: Vertebral Implant PEEK Procedure; Device: Vertebral Implant PEEK (VIP) implant

INTERVENTIONS:
Procedure: Vertebral Implant PEEK Procedure — Vertebral Implant PEEK (VIP) procedure is a minimally invasive/percutaneous vertebral augmentation (PVA), image guided procedure. Two VIP devices are implanted in each to be treated vertebra. A cavity is drilled allowing the introduction of the implant posteriorly through the pedicle and the vertebral body upto the anterior wall. A part of the implant is embedded into the pedicle, thus providing posterior support. The other part of the device, located in the vertebral body, presents a central canula and lateral perforations, which allow acrylic bone cement diffusion, filling of the vertebral body, filling and fixing the implant, and supporting of the upper endplate. The combination of the implant and the cement allows the treatment of vertebral fractures.
  Other Names: Vertebral Implant; VIP
Device: Vertebral Implant PEEK (VIP) implant — The study device is V-STRUT© Vertebral Implant manufactured by Hyprevention (VIP -Vertebral Implant PEEK), FDA cleared under K191709, indicated for use in the treatment of vertebral fractures in the thoracic and lumbar spine from T9 to L5. It is intended to be used in combination with PMMA bone cement.
  Other Names: V-STRUT©

SUMMARY:
The RECONSTRUCT study is a multi-center, prospective, single arm, post-market, pilot study to evaluate clinical and radiologic outcome data regarding the use of the Vertebral Implant PEEK (VIP) implant in the treatment of symptomatic, acute (<8week) vertebral compression fractures who have failed conservative care strategies.

DETAILED DESCRIPTION:
Vertebral compression fractures affect an estimated 1.4 million patients in the world annually and incidence rates rise exponentially with age, especially in women. Outcomes following non-interventional management of these injuries are generally poor, largely as a consequence of opioid requirements, prolonged immobilization, and bedrest. As a result, interventional techniques such as balloon kyphoplasty and vertebroplasty with or without implantable devices are currently regarded as the standard of care for select patients with acute painful osteoporotic compression fractures. These procedures relieve fracture pain by stabilizing the fracture site using cement.

Alternative interventional techniques include percutaneous vertebral augmentation, which combine cement injection with implantable devices, such as the SpineJack® and KIVA® devices. The RECONSTRUCT study will build on the outcomes of the SAKOS and KAST clinical trails that evaluated the SpineJack® and KIVA® devices, respectively.

The Vertebral Implant PEEK (VIP) implant (V-STRUT© manufactured by Hyprevention) has undergone both clinical and pre-clinical testing. Static and dynamic bending of the implant has been evaluated to demonstrate that the product is capable of supporting in-situ loading, and increase fracture load and energy to fracture.

A total of 30 eligible subjects with a diagnosis of osteoporotic fractures of the thoracolumbar spine, as confirmed by MRI scan, and who are treated with the Vertebral Implant PEEK (VIP) device will be asked to join the study. No placebo or control will be utilized during this study.

RECONSTRUCT has been designed with the intention of achieving two goals: 1) to inform the design of larger controlled clinical trials in the future and 2) to assess the safety of the study device within the patient sample.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* Osteoporotic compression fractures of the thoracolumbar spine (T1 -L5)
* Up to three levels can be fractured and treated, but at least one of the three need to be treated with V-STRUT; the level(s) to be treated with study device is at the discretion of the enrolling investigator
* Fracture age of ≤ 12 weeks as indicated by onset of pain or known antecedent traumatic event with corresponding evidence of acuity on MRI (T1 and STIR sequences) or radioisotope bone scan
* ODI ≥ 30/100 at screening visit and VAS ≥ 60 at screening visit
* Failure of conservative management strategies for compression fractures resulting in inadequately controlled pain and/or patient immobility
* Patient has failed non-operative medical therapy as defined by one of the following definitions set forth by the American College of Radiology:

  1. For a patient rendered nonambulatory as a result of pain from a VCF, pain persisting at a level that prevents ambulation despite 24 hours of analgesic therapy; or
  2. For a patient with sufficient pain from a VCF such that physical therapy is intolerable, pain persisting at that level despite 24 hours of analgesic therapy; or
  3. For a patient with pain from a VCF, unacceptable side effects such as excessive sedation, confusion, or constipation as a result of the analgesic therapy necessary to reduce pain to a tolerable level.
* Magerl classification A1.1, A1.2, A1.3, A2.1, A2.2 and A3.1 type fractures: pediculosomatic junction fractures and other fractures involving vertebral pedicles
* Appropriate pedicle diameter to receive 4.5mm, 5.5mm diameter or 6.5mm diameter implants
* ASA < 4

Exclusion Criteria:

* Patient clearly improving on conservative treatment
* Any contra-indication or allergy to implant material or cement
* Systemic infection or infection located in the spine
* Any medical condition including but not limited to anemia, coagulation disorders, fibromyalgia, algoneurodystrophy, Paget's disease, uncontrolled diabetes that would preclude the patient from having surgery or would impede the benefit of surgery
* Neurologic signs or symptoms related to the fracture or the impeding pathological fracture
* Any previous surgical treatment (material or cement) in the targeted vertebra
* Less than one third of the original vertebral body height remaining
* Unstable fractures or neoplasms with posterior involvement
* Damages of the posterior wall
* Sclerotic cancellous bone
* Pedicles not large enough to accept V-STRUT© instrumentation and implants
* Pregnancy(women of childbearing potential must have a negative pregnancy test to participate)
* Pre-existing or clinically unstable neurologic deficit
* Spinal canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level to be treated
* Any physical exam evidence of myelopathy or radiculopathy
* Pain based on clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis (progressive weakness or paralysis)
* Bedbound prior to incident fracture
* Spondylolisthesis >Grade 1 at target VB
* Any underlying systemic bone disease other than osteoporosis (e.g., osteomalacia, osteogenesis imperfect, Paget's disease, etc.)
* A medical contraindication to spinal surgery and/or general anesthesia, such as coagulopathy and/or taking warfarin (Coumadin) or other anticoagulant or anti-aggregate (anti-platelet agents) on regular basis for coagulopathy (with a threshold for normal being INR≤1.5, PTT within lab normal range, and platelet count > 100,000)
* Disabling backpain due to causes other than acute fracture
* Severe cardiopulmonary deficiencies
* Any evidence of alcohol or drug abuse
* Uncontrolled psychiatric illness or severe dementia
* Involved in medical litigation including workers' compensation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | End of study at 18 months
  Safety will be measured by number of device related serious adverse events using Common Terminology Criteria for Adverse Events (CTCAE) v4.0

SECONDARY OUTCOMES:
Procedure duration | Day 1, at end of procedure
  Procedure duration in minutes
Volume of cement injected | Day 1, at end of procedure
  volume of cement injected per level
Cement leakage | Day 1, at end of procedure
  Presence of cement leakage
Fluoroscopy time | Day 1, at end of procedure
Fluoroscopy dose | Day 1, at end of procedure
Vertebral Height | 6 months
  percentage of vertebral height restoration
Visual Analogue Symptom (VAS) | 6 months
  Pain VAS, full range from 0-100, with higher score indicating more pain
The Oswestry Disability Index | 6 months
  The Oswestry Disability Index is a Low Back Pain Disability Questionnaire frequently used to assess function and very often report in the literature. Full range from 0-100, with higher score indicating more severe disability.
Lost to follow up rate | 6 months
  Study will evaluate the lost to follow up rate to determine statistical methodology and enrollment requirements for any follow up pivotal study

CONTACTS AND LOCATIONS:
Overall Officials: Tomoyoshi Shigematsu, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Johns Hopkins, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - St. Luke's, Bethlehem, Pennsylvania
  - West Virginia, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
Upon the completion of the study, Mount Sinai's data management team will clean and analysis all data in preparation of manuscript writing and publication. The intention will be to publish together between the principal investigator and the sponsor.
  Following publication, Mount Sinai will archive and store all associated data on it's cloud-based system